CLINICAL TRIAL: NCT05068648
Title: Wheelchair Backs That Support the Spinal Curves: Assessing Postural and Functional Changes
Brief Title: Wheelchair Backs That Support the Spinal Curves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: Kessler Institute for Rehabilitation (Industry); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director of Research and Evaluation, Craig Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#1788302
Record Dates: First submitted 2021-09-14; First posted 2021-10-06 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MWC Configuration 1 (Active Comparator): standard upholstery back that promotes posterior pelvic tilt set at or below cushion level and 1" above inferior angle
  Interventions: Other: Manual Wheelchair (MWC) backrest configuration
- MWC Configuration 2 (Active Comparator): active contour back positioned with seat gap and with free scapulae
  Interventions: Other: Manual Wheelchair (MWC) backrest configuration
- MWC Configuration 3 (Active Comparator): active contour back positioned with seat gap and with blocked scapulae
  Interventions: Other: Manual Wheelchair (MWC) backrest configuration
- MWC Configuration 4 (Active Comparator): deep contour back positioned with seat gap and with free scapulae
  Interventions: Other: Manual Wheelchair (MWC) backrest configuration
- MWC Configuration 5 (Active Comparator): deep contour back positioned without seat gap and with free scapulae
  Interventions: Other: Manual Wheelchair (MWC) backrest configuration

INTERVENTIONS:
Other: Manual Wheelchair (MWC) backrest configuration — Wheelchair backrest fitting, postural and functional assessment

SUMMARY:
The overall objective of this fully powered clinical trial is to investigate if using a solid backrest on a manual wheelchair (MWC) will improve postural alignment, function and wheelchair mobility, as compared with an upholstery backrest, and to explore the impact of overall back height, contour, and seat gap when using a solid backrest in individuals with spinal cord injury (SCI).

DETAILED DESCRIPTION:
A properly fit wheelchair and seating system can have a profound impact on the daily life of people with spinal cord injury (SCI). A backrest that supports the natural spinal curves is thought to enhance posture, functional mobility, and comfort for manual wheelchair (MWC) users. In fact, therapists routinely prescribe after-market posture-backs based on clinical reasoning. However, there is little research comparing the efficacy of an after-market posture-back to the standard upholstery back, and it is becoming increasingly difficult to justify these to group insurance payers.

Based on this, investigators performed a pilot study to investigate whether there were postural and/or functional differences between using a standard upholstery WC back and an after-market solid posture-back. The results of that study have been presented at the American Congress of Rehabilitation Medicine (ACRM) annual conference in November 2019 and the Combined Sections Meeting (CSM) of the American Physical Therapy Association (APTA) in February 2020, and were also published in the Journal of Spinal Cord Medicine in 2020.

Although the results of that study demonstrated clinical relevance and statistical trends for improvements in postural alignment and functional outcomes when using a solid back, there was not enough power to establish statistical significance. It also did not evaluate the effect of backrest height and position or depth of contour in order to inform clinical practice. The overall objective of this fully powered clinical trial is to further investigate if using a solid backrest on MWC will improve postural alignment, function and wheelchair mobility, as compared with an upholstery backrest; and to explore the impact of overall back height, seat gap, and contour when using a solid backrest.

ELIGIBILITY:
Inclusion Criteria:

* Full time manual wheelchair users
* Motor complete SCI from C6-T4
* Age 18-70 at time of testing
* Time since injury > 3 month at time of testing

Exclusion Criteria:

* Weight >250 pounds
* Current pressure ulcer at time of testing
* Significant shoulder pain that precludes independent mobility at time of testing
* Insufficient range of motion to achieve neutral pelvis and spine at time of testing
* Orthopedic restrictions requiring a brace that would impact functional outcome measures
* Shoulder flexion range of motion <120 degrees at time of testing
* PSIS-to-Inferior Angle of scapula measurement less than 8 inches or greater than 16 inches
* Cognitive deficits or visual impairment that would impair ability to give informed consent or to follow simple instructions during testing
* Children, pregnant women and prisoners will not participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Pelvic Angle | Throughout study completion; average of 2 years.
Frontal Pelvic Angle | Throughout study completion; average of 2 years.

SECONDARY OUTCOMES:
Spinal Angle of Kyphosis | Throughout study completion; average of 2 years.
Frontal Sternal Angle | Throughout study completion; average of 2 years.
Vertical Forward Reach Test (VFRT) | Throughout study completion; average of 2 years.
One Stroke Push Test | Throughout study completion; average of 2 years.
Timed Forward Wheeling | Throughout study completion; average of 2 years.
Timed ramp ascent | Throughout study completion; average of 2 years.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Craig Hospital, Englewood, Colorado
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Kessler Institute for Rehabilitation, West Orange, New Jersey